CLINICAL TRIAL: NCT02718807
Title: Use of 3-D Printed Models to Improve Patient Understanding During the Informed Consent Process: A Pilot Study
Brief Title: Rapid Prototyping Models for Patient Education
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 3980
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Patient Education
Keywords: Patient Care; Education
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post-partum Women: Post-partum women following an atraumatic pregnancy.
  Interventions: Other: RP model explanation and questionnaire
- Co-Parents: Co-parents to post-partum women following an atraumatic pregnancy.
  Interventions: Other: RP model explanation and questionnaire

INTERVENTIONS:
Other: RP model explanation and questionnaire — Rapid prototyping models of anatomy will be used to demonstrate an anatomic and medical condition and participants will grade the experience on a questionnaire.

SUMMARY:
Pre-made rapid prototyping models will be used to increase patient education versus current methodologies.

DETAILED DESCRIPTION:
Post-partum women and their co-parent will have a medical condition explained to them first verbally, followed by a questionnaire, and then with the use of anatomical models created by rapid prototyping, followed by a questionnaire. The two questionnaires will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Mother
* Post-partum
* Atraumatic delivery of healthy, live infant at HMC
* Age > 18

Co-parent

* Co-parent
* Atraumatic delivery of healthy, live infant at HMC
* Age > 18

Exclusion Criteria:

* any pregnancy related issues
* fetal loss
* NICU stay > 6 hours
* Emergent cesarean section
* Post-partum hemorrhage
* Hysterectomy
* Any other condition requiring unplanned, medical intervention during labor and delivery
* Prior fetal loss or anomaly
* Inability to read or write English
* those who do not consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-partum women and respective co-parents who are greater than 18 years of age and fluent in the English language.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference in questionnaire score | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Participant Age | through study completion, an average of 1 year
Participant Education Level | through study completion, an average of 1 year
Participant Gender | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James Mooney, MD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with participants

REFERENCES:
- [Background] Kinnersley P, Phillips K, Savage K, Kelly MJ, Farrell E, Morgan B, Whistance R, Lewis V, Mann MK, Stephens BL, Blazeby J, Elwyn G, Edwards AG. Interventions to promote informed consent for patients undergoing surgical and other invasive healthcare procedures. Cochrane Database Syst Rev. 2013 Jul 6;2013(7):CD009445. doi: 10.1002/14651858.CD009445.pub2. PMID 23832767
- [Background] Farrell EH, Whistance RN, Phillips K, Morgan B, Savage K, Lewis V, Kelly M, Blazeby JM, Kinnersley P, Edwards A. Systematic review and meta-analysis of audio-visual information aids for informed consent for invasive healthcare procedures in clinical practice. Patient Educ Couns. 2014 Jan;94(1):20-32. doi: 10.1016/j.pec.2013.08.019. Epub 2013 Aug 30. PMID 24041712
- [Background] Challoner A, Erolin C. Creating pathology models from MRI data: a comparison of virtual 3D modelling and rapid prototyping techniques. J Vis Commun Med. 2013 Jun;36(1-2):11-9. doi: 10.3109/17453054.2013.790011. PMID 23641760
- [Background] Gonzalez-Cota A, Kruger GH, Raghavan P, Reynolds PI. Computational modeling and prototyping of a pediatric airway management instrument. Anesth Analg. 2010 Sep;111(3):649-52. doi: 10.1213/ANE.0b013e3181e5ea7c. Epub 2010 Jun 25. PMID 20581164
- [Background] Mankovich NJ, Cheeseman AM, Stoker NG. The display of three-dimensional anatomy with stereolithographic models. J Digit Imaging. 1990 Aug;3(3):200-3. doi: 10.1007/BF03167610. PMID 2085555
- [Background] Mori K, Yamamoto T, Oyama K, Ueno H, Nakao Y, Honma K. Modified three-dimensional skull base model with artificial dura mater, cranial nerves, and venous sinuses for training in skull base surgery: technical note. Neurol Med Chir (Tokyo). 2008 Dec;48(12):582-7; discussion 587-8. doi: 10.2176/nmc.48.582. PMID 19106500
- [Background] Miller SF, Sanz-Guerrero J, Dodde RE, Johnson DD, Bhawuk A, Gurm HS, Shih AJ. A pulsatile blood vessel system for a femoral arterial access clinical simulation model. Med Eng Phys. 2013 Oct;35(10):1518-24. doi: 10.1016/j.medengphy.2013.04.010. Epub 2013 May 18. PMID 23688608
- [Background] Noecker AM, Chen JF, Zhou Q, White RD, Kopcak MW, Arruda MJ, Duncan BW. Development of patient-specific three-dimensional pediatric cardiac models. ASAIO J. 2006 May-Jun;52(3):349-53. doi: 10.1097/01.mat.0000217962.98619.ab. PMID 16760727
- [Background] Schubert C, van Langeveld MC, Donoso LA. Innovations in 3D printing: a 3D overview from optics to organs. Br J Ophthalmol. 2014 Feb;98(2):159-61. doi: 10.1136/bjophthalmol-2013-304446. Epub 2013 Nov 28. PMID 24288392
- [Background] Starosolski ZA, Kan JH, Rosenfeld SD, Krishnamurthy R, Annapragada A. Application of 3-D printing (rapid prototyping) for creating physical models of pediatric orthopedic disorders. Pediatr Radiol. 2014 Feb;44(2):216-21. doi: 10.1007/s00247-013-2788-9. Epub 2013 Nov 8. PMID 24202430
- [Background] Suzuki M, Ogawa Y, Hagiwara A, Yamaguchi H, Ono H. Rapidly prototyped temporal bone model for otological education. ORL J Otorhinolaryngol Relat Spec. 2004;66(2):62-4. doi: 10.1159/000077796. PMID 15162002
- [Background] Zopf DA, Hollister SJ, Nelson ME, Ohye RG, Green GE. Bioresorbable airway splint created with a three-dimensional printer. N Engl J Med. 2013 May 23;368(21):2043-5. doi: 10.1056/NEJMc1206319. No abstract available. PMID 23697530